CLINICAL TRIAL: NCT07157033
Title: A Phase 1/2a, Open Label, Dose-Escalation Study to Evaluate the Safety and Efficacy of XER-001 (Amifostibe for Nasoduodenal Delivery) in Combination With Sterotactic Body Radiotherapy for Treatment of Locally-Advanced Pancreatic Adenocarcinoma
Brief Title: A Phase 1 Study to Evaluate Safety and Efficacy of XER-001 (Amifostine for Nasoduodenal Delivery) in Combination With Sterotactic Body Radiotherapy for Treatment in Patients With Locally Advanced Pancreatic Cancer.
Acronym: XER-001
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xerient Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XER-201
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-08

CONDITIONS: Locally Advanced Pancreatic Adenocarcinoma; Locally Advanced Pancreas Cancer; Locally Advanced Pancreatic Ductal Adenocarcinoma
Keywords: locally advanced pancreatic cancer; pancreatic cancer; locally advanced pancreatic adenocarcinoma; SBRT; amifostine
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- XER-001 at increasing dose levels (Experimental)
  Interventions: Drug: XER-001

INTERVENTIONS:
Drug: XER-001 — XER-001 (Amifostine for nasoduodenal delivery)

SUMMARY:
The purpose of this study is to assess the safety, tolerability and efficacy of XER-001 and identify a best dose for future studies.

DETAILED DESCRIPTION:
The primary objective of the phase 1 component of the study is to evaluate the safety, tolerability, and PK of nasoduodenal administration of XER-001 in conjunction with stereotactic body radiotherapy (SBRT) in patients with LAPC. The primary objective of the phase 2a component of the study is to evaluate safety and efficacy of combination SBRT and XER-001 with increasingly-liberalized duodenal radiation dose constraints.

ELIGIBILITY:
Inclusion Criteria:

1. Cytologic or biopsy confirmed adenocarcinoma of the pancreas
2. Disease deemed amenable to definitive treatment with SBRT by being:

   1. Locally-advanced and/or technically unresectable, as determined by a specialist pancreaticobiliary surgeon and as part of a multidisciplinary team review including of multiphase cross-sectional imaging, demonstrating: i. Greater than 180-degree tumor involvement of the superior mesenteric artery (SMA) ii. Greater than 180-degree tumor involvement of the celiac axis including major branches of the celiac axis that would render the tumor unresectable (e.g. common hepatic artery) iii. Tumor involvement of the first branch of the SMA that is not surgically reconstructible iv. Long segment involvement of the superior mesenteric vein/portal vein/hepatic artery that is not amenable to surgical reconstructible.
   2. Potentially resectable anatomically but deemed not a surgical candidate after multidisciplinary review (such as unresectable due to comorbid conditions that render.

      the risks of surgery prohibitive)
   3. Potentially resectable but the patient elects to refuse surgery and prefers to pursue SBRT, and disease is deemed eligible for SBRT
3. Primary tumor involvement abutment of the bowel is allowed, however bowel infiltration or invasion (identified endoscopically or by contrast enhanced imaging) is not allowed.
4. No distant metastatic disease either prior to or following induction systemic therapy
5. Completion of medically indicated first line systemic therapy, which may include but is not limited to regimens such as FOLFIRNOX, gemcitabine/abraxane, and similar regimens
6. Patients must be able to understand and comply with any treatment related procedures for SBRT. including breath-hold techniques or tolerance of compression belt, or other motion management strategies for SBRT delivery.
7. Age 18 years or older
8. Eastern Cooperative Group (ECOG) performance status 0, 1, or 2
9. Adequate hematologic function as indicated by:

   1. Absolute neutrophil counts >/= 1500/mm3
   2. Hemaglobin >/= 8.0 g/dL
   3. Plor current use of hepato atelet count >/= 75,000/mm3
10. No known liver disease or hepatic impairment, as well as no recent or current use of hepatotoxic drugs or substances that could compromise liver function unless a washout period has been completed. Adequate liver function as indicated by:

    1. Total bilirubin </= 1.5x upper limits of normal (per institutional laboratory reference standard)
    2. Aspartate aminotransferase (AST) and alanine aminotranferase (ALT) </= 2.5 upper limits of normal (per institutional reference standard)
11. Baseline serum calcium level >/= 8.4 mg/dL
12. No clinically significant history or presence of safety 12-lead ECG findings as judged by the investigator at screening and check-in(s), including each criterion as listed below:

    1. Normal sinus rhythm (heart rate between 40 and 100 bpm)
    2. QTcF interval </= 470 msec
    3. QRS interval </= 110 msec
    4. and PRS interval </= 220 msec Repeat measurements may be performed at the discretion of the investigator or designee
13. An understanding, ability, and willingness to fully comply with the protocol-defined schedule of assessments, procedures, and restrictions
14. Must provide written informed consent prior to the initiation of any protocol specific procedures
15. The effects of XER-001 on the developing human fetus are unknown. For this reason women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for at least six months following the last (fifth) day of radiotherapy on this study. Exceptions to this inclusion criterion are available to women who meet any of the following criteria:

    * Postmenopausal (no menses in greater than or equal to 12 consecutive months or validated by follicle stimulating hormone [FSH] levels.
    * History of hysterectomy or bilateral salpingo-oophorectomy
    * Ovarian failure (FSH and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy)
    * History of bilateral tubal ligation or another surgical sterilization procedure
16. Approved methods of birth control are as follows: hormonal contraception (I.e. birth control pills, injection, implant, transdermal patch, vaginal ring), intrauterine device (IUD), tubal ligation or hysterectomy, subject/partner post vasectomy, implantable or injectable contraceptives, and condoms with spermacide. Not engaging in sexual activity through six months following the last (fifth) day of radiotherapy on this study is an acceptable practice; however periodic abstinence, the rhytm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

For male participants on this trial, contraception is required as above dusing the study and for at least three months following the last (fifth) day of radiotherapy on this study if the have partners who can become pregnant (woman of child-bearing potential). Similarly, male participants on this trial should not donate sperm during the study and for at lease three months following the last (fifth) day of radiotherapy on this study.

Exclusion Criteria:

1. Prior radiotherapy to the upper abdomen with overlap of. the anticipated SBRT field
2. Prior radiopharmaceutical therapy
3. Prior surgical resection of the pancreatic tumor
4. Uncontrolled or active gastric or duodenal ulcer disease within 30 days of enrollment
5. Visable invasion of tumor into the bowel/stomach.duodenal lumen on endoscopic evaluation
6. Residual or ongoing grade 3+ non-hemotological toxicity from chemotherapy other than alopecia
7. Concurrent participation in another interventional clinical trial or use of another investigational agent within 30 days of study consent. Note that participation in non-interventional clinical trials (e.g. quality of life [QOL], imaging, etc) is not exclusionary
8. Uncontrolled intercurrent illness including but not limited to: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, renal failure, cardiac arrhythmia
9. Patients with history of myocardial infarction or unstable angina within 6 months prior to study enrollment
10. Patients with history of symptomatic or (CTCAE-defined) grade 3+ hypocalcemia
11. Patients with history of hypoparathyroidism
12. Patients with history of hypertension where medical providers deem that interruption of antihypertensive regimen for one week is deemed unsafe.
13. Patients with systolic blood pressure (BP) < 100 or diastolic BP < 65 at screening or baseline
14. History or presence of a disease, such as hepatic impairment or renal insufficiency, that could affect the absorption, distribution, metabolism, or elimination of the investigational product, tolerance to radiotherapy, or could affect clinical or laboratory assessments.

    Patients with an estimated glomerular filtration rate of less than 30 mL per minute are excluded from the trial. Patients with total bilirubin greater than 2.5 mg/dL are excluded from the trial unless patient has history of Gilbert's syndrome. In case of suspected or confirmed Gilbert's syndrome, bilirubin will be fractionated, and patients with direct bilirubin greater than 1.5 mg/dL will be excluded from the trial.
15. History of cardiac-related condition, which may include, but is not limited to, torsades de pointes, ventricular fibrillation, or ventricular tachycardia
16. Presence or family history (parents and siblings) of congenital lqt syndrome or any premature history of myocardial infarction considered clinically significant by the investigator or designee
17. History or presence of palpitations, unexplained syncope, shortness of breath or any other symptoms that may relate to cardiac arrhythmias
18. Any ECG evidence of physiological variants predisposing to electrical instability (eg. frequent pre-ventricular systolic beats)
19. Medical disorder that may require treatment during the study or make the subject unlikely to complete the study.
20. Inability to fast for 3 hours prior to study drug administration
21. Known history of active hepatitis B/C or active human immunodeficiency virus (HIV) not on highly-active anti-retroviral therapy for a minimum of 30 days
22. Donation or loss of more than 500 ml of whole blood within 30 days prior to screening
23. Difficulty with venous access or unstable or unwilling to undergo catheter insertion
24. Female subjects who are currently pregnant (have a positive pregnancy test), are lactating, or planning to breastfeed. Pregnant or breastfeeding women are excluded from this study because there is an unknown risk for adverse events in nursing infants secondary to treatment of the mother with amifostine, breastfeeding should be discontinued if the mother is treated with amifostine
25. An employee of the sponsor or research site personnel directly affiliated with this study or their immediate family member defined as a spouse, parent, child, or sibling, whether biological or legally adopted
26. A subject who, in the opinion of the investigator or designee, is considered unsuitable or unlikely to comply with the study protocol for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2029-07-31 (Estimated); Study Completion 2034-07-31 (Estimated)

PRIMARY OUTCOMES:
Safety Assessments [Dose Escalation] | 18 Months
  Incidence of Dose Limiting Toxicities (DLTs) in DLT-evaluable subjects
Safety Assessments [Dose Escalation] | 18 Months
  Identify the maximum tolerated dose and the RP2D
Safety Assessments [Dose escalation and Dose Expansion] | 40 months
  Number of participants with Serious Adverse Events (SAEs) graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0
Safety Assessments [Dose Escalation and Dose Expansion] | 40 Months
  Number of participants with Treatment-related Adverse Events (AEs) graded per NCI-CTCAE version 5.0
Safety Assessments [Dose Escalation and Dose Expansion] | 40 Months
  Number of participants with Treatment-Emergent AEs (TEAEs) graded per NCI-CTCAE version 5.0
Safety Assessments [Dose Escalation and Dose Expansion] | 40 Months
  Gastrointestinal toxicity related to SBRT and LAPC

SECONDARY OUTCOMES:
Antitumor Activity | 40 Months
  Local disease control at 6 months per RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Christus St. Vincent Regional Cancer Center, Santa Fe, New Mexico
  - Oncology Consultants, P.A., Houston, Texas